CLINICAL TRIAL: NCT06954688
Title: The Influence of Dry Needling for Hypertonia and Spasticity Treatment on Neuropathic Pain in Lower Extremity of Spinal Cord Injury: A Case Series Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Need for a new version of the study to assess neuropathic pain more specifically
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Revalidatieziekenhuis RevArte (Unknown)
Responsible Party: Principal Investigator, Wim Saeys, Professor, PhD, Universiteit Antwerpen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6585
Record Dates: First submitted 2025-03-31; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Neuropathic Pain; Spasticity; Dry Needling Technique; Spinal Cord Injury
Keywords: spinal cord injury; pain; spasticity; dry needling
MeSH Terms: conditions — Neuralgia; Muscle Spasticity; Spinal Cord Injuries; Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: monocentric interventional cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dry needling (Experimental): dry needling
  Interventions: Other: dry needling

INTERVENTIONS:
Other: dry needling — Dry Needling: The puncture is intramuscular and is performed with a non-beveled, filiform, solid needle, similar to those used in acupuncture, which has been shown to produce less damage at the muscle level. It does not infiltrate any substance. As many entries as necessary are made until the local twitch response (LTR) is exhausted.

SUMMARY:
Spinal cord injury is a life-changing event that places a burden on the healthcare system, including caregivers and affected individuals. Studies do not provide a conclusive incidence rate due to methodological differences. However, a trend observed in recent years is an increasing incidence among the elderly population due to falls or non-traumatic spinal cord injury.

The clinical consequences of spinal cord injury include pain and spasticity, in addition to loss of function and activity. On average, 69% of spinal cord injury patients report pain, with one-third experiencing severe pain. A similar prevalence is seen for spasticity, which is often underreported among spinal cord injury patients. Unlike pain, spasticity is considered a common symptom in chronic spinal cord injury, with at least 35% of the SCI population suffering from this sensorimotor control disorder. These two symptoms suggest a correlation, yet clear evidence is lacking.

The secondary aim of this study is to explain the mechanisms of action of Dry Needling at various levels to better determine which subgroup of spinal cord injury patients would benefit most. A targeted study could optimize the effects of such a treatment: a better understanding of the underlying mechanisms could help with patient stratification and promote a more individualized approach, taking into account the pathogenesis of spasticity and the different mechanisms that can effectively modulate it.

Additionally, this study examines the effect of the dry needling technique on hypertonia and spasticity in the spastic calf muscles of spinal cord injury patients. Research has already shown that this technique has acute effects on hypertonia and spasticity in stroke, multiple sclerosis, and Parkinson's disease. However, reliable research on spinal cord injury is lacking-currently, only a case report has investigated these effects. Therefore, this study is well-suited to build upon that case report and provide more evidence.

Furthermore, this study serves as a prospective study to observe the correlation between neuropathic pain and spasticity over time. As a pilot study, it has established a collaboration with the REVARTE rehabilitation hospital, which has a large spinal cord injury population.

The research will be conducted under the supervision of Prof. Dr. Steven Truijen (Universiteitsplein 1, 2610 Wilrijk, Belgium, steven.truijen@uantwerpen.be) and Prof. Dr. Wim Saeys (Universiteitsplein 1, 2610 Wilrijk, Belgium, wim.saeys@uantwerpen.be), organized from the University of Antwerp. During this study, no research costs will be charged to the patient, health insurance, or research environment.

Thank you in advance for your attention to our research.

DETAILED DESCRIPTION:
2.1 Primary Objectives 2.1.1. Pain Due to chronic (neuropathic) pain has been a symptom for decreasing quality of life this study will have assessments on different scales. First, the distinction of which type will be set through the International Spinal Cord Injury Pain (ISCIP) Classification, this will identify if the participant experiences acute, chronic, neuropathic or nociceptive pain. Second, the DN4 will be used for its high accuracy in SCI neuropathic pain. Third, The PainDetect Questionnaire will be included to monitor pain severity and/or its time-dependent course.

2.2 Secondary hypothesis and objectives 2.2.1. Modified Tardieu Scale for Lower extremity: The expectation of the study Is that, as already been proven in stroke population, dry needling would decrease spasticity and/or passive resistance of the ankle flexors. Therefore the MTS will be used to assess passive resistance and angle of first catch over a timespan of six treatments. This study prefers to use the TDS instead of the more common Modified Ashworth Scale for the higher sensitivity it preserves.

2.2.2. American Spinal Injury Association Impairment Scale (ASIA): As a standard assessment in the SCI follow-up to address sensory, motrocity (strength) and reflex activity, this outcome will be used to confirm correlation between neuropathic pain and or/spasticity. The latter has already been proven to correlate more with ASIA levels B and D11.

2.2.3. Two minute walk test (2MWT): Spasticity not only gives pain and discomfort in SCI population, it also affects function such as gait. To evaluate the effect on gait by decreasing the amount of spasticity, this study uses the 2MWT to evaluate the endurance of spinal cord injury patient able to walk with or without aid.

2.2.4. Spinal Cord Independence Measure (SCIM): To determine the impact on daily activities and functioning, the SCIM measures on different levels: Activities of daily living, coordination, eating, functional mobility and incontinence. An important underlying factor as pain and/or spasticity is a burden for the functionality and the well-being of the patient. By decreasing these symptoms this study ought to improve the independency of the patient, as well as the ultimate secondary objective below.

2.2.5. Quality of Life (Sci-Qol): As mentioned, the quality of life depends subjectively on the perception and confidence of the patient, which is negatively driven by pain and spasticity. By decreasing these factors, more confidence and a better perception should be seen at the end of the study. As part of the participation level assessment, the Sci-Qol questionnaire responses will provide information on the patient's health status, where higher values represent better quality of life.

3. STUDY DESIGN A mono-centric cohort study will be done in the REVARTE rehabilitation center. The primary outcome (DN4 & PainDetect) together with the tone assessments will be tested eight times, whereas the other outcomes follow the three baselines (pre and post intervention and intervention period).

4. SELECTION OF THE SUBJECT 4.1 Inclusion and Exclusion criteria All patients with an ASIA impairment scale of B, C or D are included. This study withholds complete and patients with a 'normal' score E on the ASIA impairment scale. Inclusion age will be between 18 and 85 years old. Participants are included with minimal spasticity (TDS >1). In the ankle flexors.

Exclusion criteria were patients with severe co-existent other systemic injuries, concomitant head injury and Glasgow coma scale score <15, non-cooperative patient or patients who didn't give their informed consent.

4.2 Recruitment and Data Management Plan Recruitment will be done by the doctors and physiotherapists adjunct with the study. Potential participants will be followed and screened from the intake. A second assessment will be done by the investigator to validate if the participant can be included and does not have any exclusion criteria.

All data collection will be done digitally and will be stored by means of the REDCAP software by the principal investigator.

5. INTERVENTION Dry Needling: The puncture is intramuscular and is performed with a non-beveled, filiform, solid needle, similar to those used in acupuncture, which has been shown to produce less damage at the muscle level.

It does not infiltrate any substance. As many entries as necessary are made until the local twitch response (LTR) is exhausted. The intervention will be applied once a week for a period of six weeks.

5.1. Mechanism of action The dry needling for hypertonia and spasticity has similar objectives as the myofascial dry needling technique. First it resets the cross-bridges between actine and myosine filaments within fibres due to chronic outburst of acetylcholine neurotransmitter at the neuromuscular junction. Second, by rupturing the latter (junction), less acetylcholine leakage will be seen, thus breaking the vicious circle of chronic contraction which is called a 'trigger point'. Third, by releasing the crossbridges and consequently releasing tension around the neurovascular structures, we see a domino-effect of more blood circulation, therefore more oxygen to the muscle fibres and therefore a decrease in neuropeptides, whom we know causes central and peripheral sensitisation13.

5.2 Intervention Protocol

The following muscle groups will be focused on:

* Gastrocnemius muscle: medial and lateral head
* Soleus Muscle
* Flexor Hallucis Longus muscle All muscles will be treated in supine position. However, if patients cannot tolerate these positions, alternative positions may be considered at the discretion of the treating professional. The muscles will be stimulated with repeated insertions in an attempt to evoke at least one Local Twitch Response (LTR) at each muscle location. If an LTR is not found, the therapist will continue to attempt to find an LTR at another location. The physical therapist will be using ultrasound guidance (Butterfly portable ultrasound system) to ensure safety and evade large blood vessels and nerves.

5.3 Adverse effects As an invasive treatment, dry needling has a minor risk of adverse effects during or after the treatment14.

According to a systematic review in 2020, the most common 'minor' adverse effect were bruising, bleeding and pain during dry needling, as major adverse effects are seen to be rare. To ensure locating and evading neuro-vascular structures, the dry needling treatment will be accompanied by Ultrasound guidance (Butterfly portable Ultrasound). All adverse effects will be reported and stored in a separate form on the REDCAP platform.

6. ASSESSMENTS 6.1. Pain 6.1.1. The International Spinal Cord Injury Pain (ISCIP) Classification: This classification fits as a valid assessment that is comprehensive and feasible in use for experienced as well as non-experiences clinicians and includes all types of pain related to Spinal Cord Injury.

Protocol: This classification will be used as a identifier of neuropathic pain. This will take place only in the pre-intervention and post-intervention period (screening and 1 week after intervention period).

The Classification consists of three columns which specifies hierarchically the reported pain type.

Column 1 includes the types of nociceptive pain, neuropathic pain, other pain, and unknown pain.

Column 2 includes for the neuropathic and nociceptive categories various subtypes of pains identified in previous SCI pain classifications.

Column 3 is used to specify the primary pain source at the organ level as well as the pathology, if either is known. For the other pain category, this tier is used to specify distinct recognized pain entities or syndromes which do not fulfill the criteria for nociceptive or neuropathic pain.

Protocol: The assessment will be performed before, during and after the intervention period. The questionnaire will be presented right before the intervention, one week after the end of the intervention period and mid-intervention after the fourth week). 6.1. PainDetect Questionnaire(PD-Q) : This questionnaire has been included to monitor pain severity and/or its time-dependent course17. It is a more extensive questionnaire In comparison to the DN4 Questionnaire despite having a lower sensitivity than the latter in SCI populationn16. Still, the PD-Q was chosen over the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) because of the difference between sensitivity (PD-Q 68% versus LANSS 36%).

Protocol: Similar to the DN4 questionnaire. The assessment will be performed before, during and after the intervention period. The PD-Q will be assessed right before the intervention and one week after the end of the intervention period.

6.2. Modified Tardieu Scale (ICC > 0.85, P<0.0001): Is a 6 point scale from 0 to 5 which assess spasticity or hypertonia in three different velocities.

First the passive Range Of Motion (PROM) will be tested and identified as R2 (Full range of motion achieved when muscle is at rest and tested at V1 velocity). Next, Velocity V2 will be applied (see below)to identify any catch or resistance. Last, V3 velocity follows to identify R1 (Angle of catch seen at Velocity V3, or V2 if possible). Outcome data of this assessment will be R1, R2 and the grading of muscle resistance.

6.3.ASIA scale: A standard assessment of motor, sensory and reflex loss after spinal cord injury. Then inter-rater as was intra-rater reliability are high (ICC's 0.88-0.96 and 0.98).

Protocol: The assessment will be done before the intervention period (screening) and one week after the intervention period.

6.4. Spinal Cord Independence Measure (SCIM): With a moderate to high Inter rater reliability ( 0.696-0.983), this 17-item questionnaire on a scale of 100 points will assess the participant on activity level.

Protocol: The assessment will be done before the intervention period (screening), during the intervention period once in the third week and one week after the intervention period.

6.5 Two minute walk test: The assessment is validated to be reliable in spinal cord injury (r = 0.980, p < 0.001).

Protocol: The patient will be instructed before the test's start. Patient will be instructed to cover as much distance in two minutes with or without aid. The test requires two test samples before the actual test which also will be measured. Encouragement is allowed as well as sharing the half-time of the test.

6.6 Quality of Life Questionaire(Sci-QoL): Protocol: The assessment will be done before the intervention period (screening), during the intervention period once in the third week and one week after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Spinal Cord Injury with ASIA impairment scale of B, C or D
* Age between 18 and 85 years
* Minimal spasticity (TDS >1) in the ankle flexors.

Exclusion Criteria:

* ASIA impairment scale A or E
* severe co-existent other systemic injuries
* concomitant head injury
* Glasgow coma scale score <15
* non-cooperative patient
* No informed consent given

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
DN4 Questionnaire: | At week 1(beginning of the study, pre-intervention period) , week 4 (mid-study) and week 8 (end of the study, post-intervention period)
  This questionnaire consists of ten items (four questions) on a total score of ten points. It has a cut-off of four points to identify the reported pain as neuropathic. The DN4 Questionnaire has been identified as a reliable and sensitive assessment for neuropathic pain
PainDetect Questionnaire(PD-Q) | At week 1(beginning of the study, pre-intervention period) , week 4 (mid-study) and week 8 (end of the study, post-intervention period)
  This questionnaire has been included to monitor pain severity and/or its time-dependent course17. It is a more extensive questionnaire In comparison to the DN4 Questionnaire despite having a lower sensitivity than the latter in SCI populationn16. Still, the PD-Q was chosen over the Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) because of the difference between sensitivity (PD-Q 68% versus LANSS 36%).
The International Spinal Cord Injury Pain (ISCIP) Classification: | Twice: Pre-intervention period (week 1) and post-intervention period (week 8)
  This classification fits as a valid assessment that is comprehensive and feasible in use for experienced as well as non-experiences clinicians and includes all types of pain related to Spinal Cord Injury.

SECONDARY OUTCOMES:
Modified Tardieu Scale | Every week (week1 to week 8)
  Is a 6 point scale from 0 to 5 which assess spasticity or hypertonia in three different velocities19. First the passive Range Of Motion (PROM) will be tested and identified as R2 (Full range of motion achieved when muscle is at rest and tested at V1 velocity). Next, Velocity V2 will be applied (see below) to identify any catch or resistance. Last, V3 velocity follows to identify R1 (Angle of catch seen at Velocity V3, or V2 if possible). Outcome data of this assessment will be R1, R2 and the grading of muscle resistance.
ASIA scale | Twice: Pre-intervention period (week 1) and post-intervention period (week 8)
  A standard assessment of motor, sensory and reflex loss after spinal cord injury. The inter-rater as was intra-rater reliability are high (ICC's 0.88-0.96 and 0.98)
Spinal Cord Independence Measure (SCIM) | At week 1(beginning of the study, pre-intervention period) , week 4 (mid-study) and week 8 (end of the study, post-intervention period)
  With a moderate to high Inter rater reliability ( 0.696- 0.983), this 17-item questionnaire on a scale of 100 points will assess the participant on activity level
Two minute walk test | At week 1(beginning of the study, pre-intervention period) , week 4 (mid-study) and week 8 (end of the study, post-intervention period)
  The assessment is validated to be reliable in spinal cord injury (r = 0.980, p < 0.001). The patient will be instructed before the test's start. Patient will be instructed to cover as much distance in two minutes with or without aid. The test requires two test samples before the actual test which also will be measured. Encouragement is allowed as well as sharing the half-time of the test. This test only applies for patients able/willing to walk.
Quality of Life Questionaire(Sci-QoL) | At week 1(beginning of the study, pre-intervention period) , week 4 (mid-study) and week 8 (end of the study, post-intervention period)
  The assessment will be done before the intervention period (screening), during the intervention period once in the third week and one week after the intervention period. Specific for SCI population.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation sciences and physiotherapy (MOVANT), Antwerp, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Data is stored on the online data storage and colllection database (REDCAP). Database is available for institutions writing a formal letter to our contact person. This change in GDPR informed consent description will be asked to the participated patients to share demanded data.